CLINICAL TRIAL: NCT06889363
Title: Clinical and Radiographic Evaluation of Indirect Pulp Capping Using Platelet Rich Fibrin Versus Mineral Trioxide Aggregate in Deep Carious Molars: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Mohamed Monir Mahmoud Ahmed, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SALMA.MOHAMED.MONIR.PhD
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Dental Caries; Pulp Caping; Indirect Pulp Treatment; Indirect Pulp Cap; Indirect Pulp Capping; Indirect Pulp Therapy; Deep Carious Lesion; Deep Carious Lesions; Molar Caries; Carious Molars
Keywords: Molar caries; MTA; PRF; Indirect pulp capping; Deep carious lesion; carious molars; platelet rich fibrin
MeSH Terms: conditions — Dental Caries | interventions — Pemetrexed; mineral trioxide aggregate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deep carious molars, indirect pulp capping using PRF then GI base then composite restoration (Experimental): Deep carious molars, indirect pulp capping using PRF then GI base then composite restoration
  Interventions: Biological: PRF
- Deep carious molars, indirect pulp capping using MTA then GI base then composite restoration (Active Comparator): Deep carious molars, indirect pulp capping using MTA then GI base then composite restoration
  Interventions: Drug: MTA

INTERVENTIONS:
Drug: MTA — The indirect pulp capping will be applied using MTA using an MTA carrier, then glass ionomer will be applied, then composite restoration above
  Other Names: mineral trioxide aggregate
  Arms: Deep carious molars, indirect pulp capping using MTA then GI base then composite restoration
Biological: PRF — The indirect pulp capping will be applied using PRF on a membrane, then glass ionomer will be applied , then composite restoration above
  Other Names: platelet rich fibrin
  Arms: Deep carious molars, indirect pulp capping using PRF then GI base then composite restoration

SUMMARY:
The aim of this study is the clinical and radiographic evaluation of (Platelet-Rich Fibrin (PRF) versus Mineral Trioxide Aggregate (MTA) in indirect pulp capping when used with deep carious molars over 1 year follow up.

DETAILED DESCRIPTION:
-PICOTS : P: Asymptomatic deep carious molars. I: Indirect pulp capping using PRF. C: Indirect pulp capping using MTA.

O:

Outcome name Measuring device Measuring unit

Primary outcome:

clinical findings : Pulp sensibility using cold test (Sharma A et al., 2020).

Secondary outcome:

Radiographic findings :Dentin bridge measurement in mm using digital radiographic ruler Digital Periapical using paralleling technique (Sharma A et al., 2020).

T:

T0: Baseline T1: 3 months T2: 6 months T3: 12 months S: Randomized clinical trial.

- Research question: Will PRF provide comparable clinical and radiographic outcomes to MTA in indirect pulp capping when used in deep carious molars?

ELIGIBILITY:
Inclusion Criteria:

* o Patients with asymptomatic deep carious molars.

  * Patients with clinically and radiographically confirmed deep carious lesions that do not exhibit spontaneous pain.
  * Permanent molars only.
  * Teeth with intact or minimally restored occlusal surfaces (i.e., no extensive restorations or fractures).
  * No history of previous endodontic treatment or direct pulp capping on the study tooth.
  * No signs of periapical pathology based on radiographic evaluation.
  * Patients willing to participate and follow up for 12 months.
  * Patients who agree to return for scheduled follow-ups at 3, 6, and 12 months.

Exclusion Criteria:

* o Patients with systemic conditions affecting bone or tissue healing (e.g., uncontrolled diabetes, osteoporosis, immunosuppressed conditions).

  * Pregnant or lactating women (if applicable to your study).
  * Teeth with pulp exposure or necrotic pulp.
  * Presence of symptomatic irreversible pulpitis (e.g., spontaneous pain, lingering pain).
  * Periapical pathology or internal/external resorption detected radiographically.
  * Severely broken down or non-restorable teeth.
  * Calcified root canals or excessive sclerosis that could affect pulp testing reliability.
  * Any pre-existing root canal treatment on the selected tooth.
  * Patients who have undergone recent fluoride treatment, pulpotomy, or other pulp therapies in the past 6 months.
  * Patients using medications affecting bone and tissue regeneration (e.g., bisphosphonates, corticosteroids).
  * Patients unwilling or unable to commit to the 12-month follow-up schedule.
  * Patients with poor oral hygiene or high caries risk that could compromise treatment outcomes.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pulp sensibility using cold test | baseline, 3 , 6, 12 months
  clinical finding of the investigated tooth measured with binary (yes or no)

SECONDARY OUTCOMES:
Radiographic finding | baseline, 3 , 6, 12 months
  Digital Periapical using paralleling technique (Dentin bridge measurement in mm using digital radiographic ruler)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, القاهرة - Cairo Governorate, Egypt